CLINICAL TRIAL: NCT02994186
Title: Longitudinal Assessment of Cognitive Function Following Bariatric Surgery or Medical Weight Loss Treatment
Brief Title: Examination of Cognitive Function in Obesity and Following Weight Loss
Status: Withdrawn | Type: Observational
Why Stopped: funding
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Lumos Labs, Inc. (Industry)
Responsible Party: Principal Investigator, Vance L. Albaugh, MD, PhD, Postdoctoral Fellow and Resident Surgeon, Vanderbilt University Medical Center
Other Study IDs: 161918
Record Dates: First submitted 2016-12-12; First posted 2016-12-15 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Obesity; Bariatric Surgery Candidate; Weight Loss
Keywords: cognitive function; obesity; bariatric surgery; metabolic surgery
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Surgical Weight Loss: Patients in this group are those that will be undergoing bariatric surgery (either Roux-en-Y gastric bypass or vertical sleeve gastrectomy).
  Interventions: Procedure: Bariatric Surgery
- Medical Weight Loss: Patients in this group are those who are being enrolled in a supervised medical weight loss program.
  Interventions: Other: Medical Weight Loss Program

INTERVENTIONS:
Procedure: Bariatric Surgery — These are patients who will be having either Vertical Sleeve Gastrectomy or Roux-en-Y Gastric Bypass.
  Groups: Surgical Weight Loss
Other: Medical Weight Loss Program — These are patients who will be starting a structured medical weight loss program.
  Groups: Medical Weight Loss

SUMMARY:
Bariatric surgery is the most effective, long-term treatment for morbid obesity, and consistent with previous findings, individuals who lose significant weight after surgery also have improved cognition or "brain function". The mechanisms behind these cognitive improvements are currently unknown, but are the focus of much research effort. The goal of this pilot study is to thoroughly describe these changes in surgical versus medical weight loss patients over time in a repeated measures fashion.

DETAILED DESCRIPTION:
Recent studies have demonstrated that obesity is associated with decreased cognitive function and, interestingly, weight loss is associated with improved cognitive function. Bariatric surgery is the most effective, long-term treatment for morbid obesity, and consistent with these previous findings, individuals who lose significant weight after surgery appear to have improved cognition. Previous results have only reported the appearance of cognitive improvements starting at three months postoperatively, thus, the main focus of this study is to discover whether cognitive function improvements are seen as early as one month after bariatric surgery. An acceleration in the onset of cognitive function changes could provide insight towards the ambiguous underlying neural mechanisms. The benefits of bariatric surgery extend beyond reversible cognitive deficits. Many of the medical comorbid conditions that these patients have before surgery (e.g. high blood pressure, high cholesterol, diabetes) typically resolve prior to any significant weight loss. The mechanisms for these weight-independent improvements are also undetermined. A secondary focus of this study is to determine whether or not cognitive function following bariatric surgery also improves prior to significant weight loss. To test whether cognitive function changes following bariatric surgery, two cohorts of surgical patients will be recruited as well as another group of patients undergoing medical weight loss treatment. The goal of this pilot study is to reproduce and expand upon previous findings that demonstrate cognitive improvements following bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Within the age rage of 18-70 years
* Able to give informed consent

Exclusion Criteria:

* Neurological disorder or previous injury (e.g. stoke, dementia, seizures, traumatic brain injury)
* History of any moderate to severe head injury (i.e. >5 minutes of loss of consciousness)
* History of severe psychiatric illness requiring current pharmacologic therapy(e.g. schizophrenia, bipolar disorder, personality disorders)
* History of illicit drug or alcohol abuse
* Known diagnosis of learning or developmental disability
* Impaired sensory function
* Any prior suicide attempt
* Revisional bariatric surgery
* Current or former tobacco user / smoker
* Currently pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that will be recruited for this study are those individuals that are pursuing either medical or surgical weight loss options at the Vanderbilt Centers for Medical and Surgical Weight Loss.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Cognitive Function Score | Repeated Measures Up to 6 Months
  Within group and between group longitudinal measurements will be made using longitudinal regression methods. Baseline as well as 1, 3 and 6 month measurements will be captured either from the time of bariatric surgery or initiation of a supervised medical weight loss program.
Cognitive Function Score - Surgical Group Comparison | Repeated Measures Up to 6 Months
  Within group and between group longitudinal measurements will be made using longitudinal regression methods. Baseline as well as 1, 3 and 6 month measurements will be captured either from the time of bariatric surgery or initiation of a supervised medical weight loss program. The bariatric operation will be included (Roux-en-Y gastric bypass vs. Vertical Sleeve Gastrectomy) as a variable in the regression model for between and within subjects comparisons in the bariatric surgery group.

SECONDARY OUTCOMES:
Cognitive Function Score - Crossover Patients | Repeated Measures Up to 6 Months
  There will be a group of patients that will crossover at 6 months from the medical weight loss group to the surgical weight loss group. The cognitive function score in these patients will be compared between treatment groups, as they will effectively be represented in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Vance L Albaugh, MD, PhD, Principal Investigator — Vanderbilt University Medical Center; Naji N Abumrad, MD, Study Director — Vanderbilt University Medical Center

IPD SHARING:
Plan to Share IPD: No